CLINICAL TRIAL: NCT05324774
Title: Phase III Clinical Study of the Efficacy and Safety of 9MW0813 and Aflibercept (EYLEA®) in Patients With Diabetic Macular Edema (DME) in a Multicenter, Randomized, Double-blind, Parallel Active-controlled Study
Brief Title: Efficacy and Safety of 9MW0813 in Subjects With Diabetic Macular Edema
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9MW0813-2021-CP301
Record Dates: First submitted 2022-03-30; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Macular Edema
Keywords: aflibercept; biosimilarity
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW0813 (Experimental)
  Interventions: Drug: 9MW0813
- aflibercept (Active Comparator)
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: 9MW0813 — The active ingredient of 9MW0813 injection is recombinant human vascular endothelial growth factor receptor-antibody fusion protein.
  9 doses(2mg) of the drug will be injected intravitreously.
  Arms: 9MW0813
Drug: Aflibercept — Aflibercept (trade name: Eylea®/EYLEA®) is an anti-VEGF drug developed by Regeneron/Bayer. It is a fusion protein of human VEGFR1 and VEGFR2 extracellular domains and human immunoglobulin Fc segment genes.
  9 doses(2mg) of the drug will be injected intravitreously.
  Other Names: Eylea®
  Arms: aflibercept

SUMMARY:
Phase III clinical study of the efficacy and safety of 9MW0813 and aflibercept (EYLEA®) in patients with diabetic macular edema (DME) in a multicenter, randomized, double-blind, parallel active-controlled study.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, parallel controlled phase 3 clinical trial.

The primary objective is to compare the similarity of clinical efficacy of intravitreal 9MW0813 injection and aflibercept intraocular injection (EYLEA®) in DME patients.

The secondary objectives are to compare the similarity of safety, immunogenicity and pharmacokinetics of intravitreal 9MW0813 injection and aflibercept intraocular injection (EYLEA®) in DME patients.

ELIGIBILITY:
Main Inclusion Criteria:

1. Age ≥ 18 years old, gender is not limited;
2. Diagnosed with type 1 or type 2 diabetes, and HbA1c≤10.0%;
3. The visual impairment of the study eye was mainly caused by diabetic macular edema;
4. OCT examination at screening and baseline, diabetic macular edema involving the fovea of the study eye, and central retinal thickness (CRT) ≥ 300 μm (using SD-OCT);
5. The best-corrected visual acuity (BCVA) of the study eye at screening and baseline measured using the Early Treatment of Diabetic Retinopathy Study (ETDRS) chart was between 73 and 24 letters (inclusive) (approximately equivalent to Snellen's visual acuity) score 20/40 to 20/320).

Main Exclusion Criteria:

1. Active proliferative diabetic retinopathy (PDR) exists in the study eye;
2. Structural damage to the fovea in the study eye, which may not improve BCVA after resolution of macular edema (eg, retinal pigment epithelial cell atrophy, subretinal fibrosis or scarring, significant macular ischemia, or organizing hard exudates) );
3. The study eye has any ocular disease or past medical history other than diabetic macular edema, and the investigator believes that it may affect the macular assessment or central vision (such as: cataract, retinal vascular occlusion, retinal detachment, macular traction, macular epiretinal membrane , macular hole, macular hemorrhage, preretinal fibrous proliferation involving the macula, various choroidal neovascularization);
4. The study eye has erythema of the iris, vitreous hemorrhage or traction retinal detachment;
5. The study eye has poorly controlled glaucoma (defined as intraocular pressure ≥25mmHg after anti-glaucoma drug treatment);
6. The study eye has received or may have received glaucoma filtration surgery (such as: trabeculectomy, sclerectomy and non-penetrating trabecular surgery) during the study period;
7. The study eye has received vitreoretinal surgery in the past;
8. Aphakic (except intraocular lens) in the research eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Best Corrected Visual Acuity (BCVA) | 8 weeks
  Change from Baseline in BCVA as measured by Early Treatment Diabetic Retinopathy Study(ETDRS) letter score
Change from Baseline in Central Retinal Thickness（CRT） | 8 weeks
  Change from Baseline in CRT as measured by optical coherence tomography

SECONDARY OUTCOMES:
Incidence of adverse events | 52 weeks
Immunogenicity of IVT injection of 9MW0813 and aflibercept | 52 weeks
  Anti-drug antibody (ADA) in serum is detected, ADA-positive samples will be subjected to titer analysis and neutralizing antibody (Nab) analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing tongren hospital affliated to capital medical university, Beijing, Beijing Municipality, China